CLINICAL TRIAL: NCT02988674
Title: Prospective, Multi-Center, Observational, Program to Assess Retention Rate, Persistence and Adherence in Population of Spondylarthritis (Ankylosing Spondylitis and Psoriatic Arthritis) Patients Treated With Adalimumab in Routine Clinical Settings in Russian Federation
Brief Title: A Study to Assess Retention Rate, Persistence and Adherence in Population of Spondylarthritis (Ankylosing Spondylitis and Psoriatic Arthritis) Patients Treated With Adalimumab in Routine Clinical Settings in Russian Federation
Acronym: Adherence
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-672
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Spondylarthritis; Psoriatic Arthritis; Ankylosing Spondylitis (AS)
Keywords: Adalimumab; Ankylosing spondylitis; Psoriatic arthritis; Spondylarthritis; Humira®
MeSH Terms: conditions — Spondylarthritis; Arthritis, Psoriatic; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Spondylarthritis: Participants with Spondylarthritis (ankylosing spondylitis and psoriatic arthritis) treated with adalimumab in routine clinical settings in the Russian Federation.

SUMMARY:
The objective of this study is to access retention rate, persistence and adherence in population of spondylarthritis (SpA) (ankylosing spondylitis (AS) and psoriatic arthritis (PsA)) participants treated with adalimumab in routine clinical settings in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AS or PsA.
* Planned prescription or prescribed no more than 1 month before to enrolment therapy with adalimumab. Treatment has to be prescribed according to the local product label and prescription guidelines.
* At the moment of start of treatment with adalimumab moderate/severe AS or PsA (BASDAI > 4 for AS; DAS28 >3,2 for PsA).
* Negative result of tuberculosis (TB) screening test and TB specialist permission to start biologic therapy.
* Authorization (Consent) for Use/Disclosure of Data signed by the participant.

Exclusion Criteria:

* Has contraindications for the treatment with adalimumab (please see the latest version of the locally approved label).
* Participants who are unable to walk and perform basic self-care activities either due to SpA or a comorbid condition.
* Any biologic drugs taken over before 3 months of enrolment to the study.
* Previous participation in this program.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spondylarthritis (ankylosing spondylitis and psoriatic arthritis) participants treated with adalimumab in routine clinical settings in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Proportion of participants on adalimumab therapy | Up to 30 days after administering last dose in the study (52 weeks)
  This is used to assess retention rate. Persistence/Adherence of SpA patient to treatment, as well as retention rate, is an important factor of achieving of treatment goals. Medical non-adherence poses a significant limitation to treating to target in RA and SpA.
Number of participants on adalimumab therapy | Up to 30 days after administering last dose in the study (52 weeks)
  This is used to assess retention rate. Persistence/Adherence of SpA patient to treatment, as well as retention rate, is an important factor of achieving of treatment goals. Medical non-adherence poses a significant limitation to treating to target in rheumatoid arthritis (RA) and SpA.

SECONDARY OUTCOMES:
Assessing medication persistence | Up to 48 weeks of treatment period
  Medication persistence is defined as the duration of time from initiation to discontinuation of therapy.
Assessing medication adherence | Up to 48 weeks of treatment period
  Medication adherence is defined as the extent to which a participant acts in accordance with the prescribed interval and dose of a dosing.
Change of disease activity in participants with PsA | Up to 48 weeks of treatment period
  This is assessed using Disease activity score 28 joints count (DAS28) in participants with PsA.
Change of disease activity in participants with AS | Up to 48 weeks of treatment period
  This is assessed using Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in participants with AS.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (14):
- Russia (14):
  - Kemerovo Regional Clinical Hospital n.a. S.V. Belyaev /ID# 167025, Kemerovo, Kemerovo Oblast
  - Clinical Hospital No.1 n.a. N.I.Pirogov /ID# 154379, Moscow, Moscow
  - Ivanovo Regional Clinical Hosp /ID# 167028, Ivanovo
  - Institution KhMAO-Ugra /ID# 154381, Khanty-Mansiysk
  - State Clinical policlinic /ID# 154374, Moscow
  - Central Research Institute /ID# 154375, Moscow
  - Research Institute of Rheum /ID# 154378, Moscow
  - Advisory-diagnostic Hospital /ID# 154382, Moscow
  - State Clinical Hospital /ID# 154373, Moscow
  - GBUZ Republican Hospital /ID# 167029, Petrozavodsk
  - Nort-Western State Medical Uni /ID# 154376, Saint Petersburg
  - Smolensk station JSC Russian R /ID# 167027, Smolensk
  - Tula Regional Clinical Hospita /ID# 155539, Tula
  - Yaroslavi State Medical Univer /ID# 154383, Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-672.pdf